CLINICAL TRIAL: NCT07024706
Title: The MAVRiC Study: A Phase II Study of Disease Risk Mutation Guided Finite Duration Acalabrutinib Plus Venetoclax for Relapse in CLL/SLL After First-line Finite Covalent BTKi Plus BCL2i Combination, With or Without Obinutuzumab
Brief Title: Phase 2 Study of Disease Risk Mutation-Guided Finite Acalabrutinib+Venetoclax for Relapsed CLL Post-1L Finite cBTKi+BCL2i ± Obinutuzumab
Acronym: MAVRiC
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: AbbVie (Industry); Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D8220C00036
Record Dates: First submitted 2025-05-26; First posted 2025-06-17 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Chronic Lymphocytic Leukemia (CLL); Small Lymphocytic Lymphoma (SLL)
Keywords: Chronic Lymphocytic Leukemia (CLL); Small Lymphocytic Lymphoma (SLL); Relapsed CLL; Refractory CLL; Acalabrutinib
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell | interventions — acalabrutinib; venetoclax

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Acalabrutinib and Venetoclax (Experimental): For Cohort 1, each participant will be in the study for approximately 5 years (60 months) counting from C1D1, starting with 2 cycles of acalabrutinib lead-in treatment, followed by 12 cycles of AV combination treatment, and 4 years of follow-up.
  For Cohort 2, each participant will be in the study for approximately 5 years (60 months) counting from C1D1 starting with 2 cycles of acalabrutinib lead-in treatment, followed by 22 cycles of AV combination treatment, and 3 years of follow-up.
  Interventions: Drug: Acalabrutinib; Drug: Venetoclax

INTERVENTIONS:
Drug: Acalabrutinib — Acalabrutinib is an orally available cBTKi that inhibits the activity of BTK and prevents the activation of the B-cell antigen receptor (BCR) signaling pathway.
  Other Names: CALQUENCE®
Drug: Venetoclax — Venetoclax is an orally bioavailable inhibitor of the anti-apoptotic protein BCL-2
  Other Names: Venclexta®; Venclyxto®

SUMMARY:
This study will evaluate the efficacy and safety of finite-duration acalabrutinib plus venetoclax therapy in patients with relapsed CLL or SLL, and have previously responded to first line (1L) cBTKi + BCL2i therapy (± obinutuzumab) and maintained a response for at least two years post-treatment.

DETAILED DESCRIPTION:
The purpose of this study is to explore the use of second line (2L) treatment with AV after relapse following first line (1L) cBTKi + BCL2i by assessment of ORR in participants with CLL/SLL. This study will generate efficacy and safety data needed to understand outcomes associated with AV in patients who initially responded with partial remission (PR) or better for a minimum of 2 years from the end of 1L cBTKi + BCL2i combination treatment and are experiencing clinical relapse requiring further treatment. MAVRiC explores AV as second-line (2L) CLL/SLL treatment after relapse on first-line (1L) cBTKi + BCL-2 by assessment of overall response rate (ORR)

* The study duration for each participant will be up to 5 year.
* The study consists of screening, treatment, and post-intervention follow-up periods.
* Participants will be grouped into low or high risk cohorts based on disease risk determined by IGHV mutation and TP53 aberrancy.

ELIGIBILITY:
Main Inclusion Criteria:

1. Participant must be ≥ 18 years at the time of signing informed consent.
2. Diagnosis of CLL/SLL according to iwCLL guidelines 2018 (Hallek et al. 2018)
3. Participants must have received first line treatment with fixed duration covalent BTKi plus BCL2i therapy (± obinutuzumab) with a response ≥ PR (i.e., CR, CRi, nPR, or PR) with a minimum of 2 years since the end of the prior 1L treatment.
4. The following data must be available or at least the appropriate samples drawn/acquired prior to dosing:

   1. IGHV (mutated vs. unmutated)
   2. del(17p) (present or absent)
   3. TP53 mutation (present or absent)
5. ECOG performance status 0, 1 or 2
6. Adequate organ and bone marrow (BM) function.

Main Exclusion Criteria:

1. Any evidence of diseases that, in the investigator's opinion, makes it undesirable for patient to participate in the study.
2. Significant cardiovascular or cerebrovascular disease.
3. Active bleeding or history of bleeding diathesis (e.g., hemophilia or von Willebrand disease).
4. Child-Pugh B/C liver cirrhosis.
5. History of prior or current malignancy.
6. HIV positive
7. History of progressive multifocal leukoencephalopathy (PML).
8. Active hepatitis B or C infection:
9. Corticosteroid use > 20 mg within 1 week before the first dose of study intervention.
10. History of hypersensitivity or anaphylaxis to study intervention(s).
11. Requires treatment with a strong CYP3A4 inhibitor/inducer.
12. Requires or receiving anticoagulation with warfarin or equivalent vitamin K antagonists.
13. Major surgical procedure within 30 days of the first dose of study intervention.

Ages: 18 Years to 130 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2026-01-30 (Estimated); Primary Completion 2029-05-01 (Estimated); Study Completion 2029-05-15 (Estimated)

PRIMARY OUTCOMES:
Overall Response Rate (ORR) | ORR assessed at multiple timepoints during treatment period (each cycle is 28 days). Timepoint for primary analysis is at completion of cycle 14
  ORR, defined as the proportion of participants who achieve best response of CR, CRi, nPR, or PR per iwCLL criteria as assessed by the investigator.

SECONDARY OUTCOMES:
Progression Free Survival (PFS) | PFS will be assessed from Cycle 3 to Cycle 24 during treatment period (each cycle is 28 days)
  PFS is defined as time from date of the first dose until progression per iwCLL criteria or death due to any cause in the absence of progression.
Duration of Response (DoR) | DoR will be assessed from Cycle 3 to Cycle 24 during treatment period (each cycle is 28 days)
  DoR is defined as the time from the date of first documented response until date of documented progression per iwCLL criteria or death due to any cause.
Event Free Survival (EFS) | EFS will be assessed from Cycle 3 to Cycle 24 during treatment period (each cycle is 28 days)
  EFS is defined as the time from date of the first dose until the first occurrence of disease progression, initiation of subsequent CLL/SLL therapy, or death due to any cause.
Time to Next Treatment (TTNT) | TTNT will be assessed from Cycle 3 to Cycle 24 during treatment period (each cycle is 28 days)
  TTNT is defined as the time from date of the first dose to the initiation of subsequent CLL/SLL therapy or death due to any cause
Overall Survival (OS) | OS will be assessed every 3 months through the study completion, for 5 years
  OS is defined as the time from date of the first dose until the date of death due to any cause.
Rate of undetectable Minimal Residual Disease (uMRD) | uMRD will be measured at 3 months after last treatment
  Rate of peripheral blood (PB) uMRD, defined as proportion of participants achieving remission based on a clonoSEQ® assay result of <1 CLL cell per 100,000 leukocytes (< 10-5).
Treatment-Emergent Adverse Events (safety and tolerability) of second-line (2L) treatment with Acalabrutinib and Venetoclax after relapse following 1L cBTKi + BCL2i | Safety and tolerability will be evaluated throughout the study for 5 years
  Safety and tolerability will be evaluated in terms of AEs/SAEs, AEs leading to treatment discontinuation and deaths, and relevant clinical laboratory results.

CONTACTS AND LOCATIONS:
Locations (24):
- United States (3):
  - Research Site, Boston, Massachusetts
  - Research Site, Charlotte, North Carolina
  - Research Site, Durham, North Carolina
- Research Site, Horn, Austria
- Czechia (3):
  - Research Site, Brno
  - Research Site, Hradec Kralova
  - Research Site, Ostrava
- Research Site, Dublin, Ireland
- Italy (7):
  - Research Site, Lugo
  - Research Site, Meldola
  - Research Site, Milan
  - Research Site, Padua
  - Research Site, Roma
  - Research Site, Rome
  - Research Site, Torino
- Poland (5):
  - Research Site, Bydgoszcz
  - Research Site, Krakow
  - Research Site, Lodz
  - Research Site, Lublin
  - Research Site, Warsaw
- Spain (4):
  - Research Site, Barcelona
  - Research Site, Granada
  - Research Site, Madrid
  - Research Site, Majadahonda

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All requests will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the de-identified individual patient-level data in an approved sponsored tool. Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information.
URL: https://vivli.org/